CLINICAL TRIAL: NCT01618695
Title: A Double-blind, Placebo-controlled, Parallel-group Study With an Open-label Extension Phase to Evaluate the Efficacy and Safety of Perampanel (E2007) Administered as an Adjunctive Therapy in Subjects With Refractory Partial-onset Seizures
Brief Title: A Study With an Open-label Extension Phase to Evaluate the Efficacy and Safety of Perampanel (E2007) Administered as an Adjunctive Therapy in Subjects With Refractory Partial-onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2007-J000-335
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Results first posted 2020-06-05 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Partial-onset Seizures
Keywords: Partial-onset Seizures; partial seizures; seizure; epilepsy
MeSH Terms: conditions — Seizures; Epilepsy | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perampanel (Experimental)
  Interventions: Drug: Perampanel
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Perampanel — Core study: 4 milligram (mg) group- Week 0 Once daily 2 milligram per day (mg/day), Week 1 to Week 18 Once daily 4 mg/day; 8 mg group- Week 0 Once daily 2 mg/day, Week 1 Once daily 4 mg/day, Week 2 Once daily 6 mg/day, Week 3 to Week 18 Once daily 8 mg/day; 12 mg group- Week 0 Once daily 2 mg/day, Week 1 Once daily 4 mg/day, Week 2 Once daily 6 mg/day, Week 3 Once daily 8 mg/day, Week 4 Once daily 10 mg/day, Week 5 to Week 18 Once daily 12 mg/day.
  Extension study: 4 mg group- Week 19 to Week 22 Once daily 4 mg/day, Week 23 Once daily 6 mg/day, Week 24 Once daily 8 mg/day, Week 25 Once daily 10 mg/day, Week 26 to Week 75 or more Once daily 12 mg/day; 8 mg group- Week 19 to Week 22 Once daily 8 mg/day, Week 23 Once daily 10 mg/day, Week 24 to Week 75 or more Once daily 12 mg/day; 12 mg group- Week 19 to Week 75 or more Once daily 12 mg/day.
  Other Names: E2007
  Arms: Perampanel
Drug: Placebo — Core study: Week 0 to Week 18 Once daily placebo.
  Extension study:
  Week 19 to Week 22 Once daily placebo, Week 23 Once daily perampanel 2 mg/day, Week 24 Once daily perampanel 4 mg/day, Week 25 Once daily perampanel 6 mg/day, Week 26 Once daily perampanel 8 mg/day, Week 27 Once daily perampanel 10 mg/day, Week 28 to Week 75 or more Once daily perampanel 12 mg/day.
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm the efficacy and safety of perampanel compared to placebo in patients with refractory partial-onset seizures

ELIGIBILITY:
Inclusion Criteria

1. Male or female and greater than or equal to 12 years of age;
2. Have a diagnosis of epilepsy with partial seizures with or without secondarily generalized seizures
3. Participants with computed tomography (CT) or magnetic resonance imaging (MRI) diagnosis within the last 10 years (for adults) and 5 years (for adolescents) prior to visit 1 that ruled out progressive central nervous system (CNS) disorders, example, neurodegenerative disorders, brain tumors. For participants without existing CT or MRI results, CT or MRI was performed at or after Visit 1 but results evaluation was performed by Visit 2
4. Participants who had been treated for at least 12 weeks but confirmed to be uncontrolled with more than one standard antiepileptic drug (AED) for 2 years before enrollment
5. During the 6-week Prerandomization Phase participants must have had greater than or equal to 5 partial seizures per 6-week
6. Are currently being treated with stable doses and administrations of 1, 2, or a maximum of 3 approved AEDs. Only 1 inducer AED (defined as carbamazepine, phenytoin or oxcarbazepine only) out of the maximum of 3 AEDs is allowed

Exclusion Criteria

1. Presence of nonmotor simple partial seizures only;
2. Presence of primary generalized epilepsies or seizures, such as absences and/or myoclonic epilepsies;
3. Presence or previous history of Lennox-Gastaut syndrome;
4. A history of status epilepticus within 1 year prior to screening
5. Seizure clusters where individual seizures cannot be counted
6. A history of psychogenic seizures within 5 years prior to screening

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 940 (Actual)
Dates: Start 2012-05-15 (Actual); Primary Completion 2014-09-15 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (117):
- Australia (7):
  - Facility #1, Bedford Park
  - Facility #1, Camperdown
  - Facility #1, Clayton
  - Facility #1, Fitzroy
  - Facility #1, Heidelberg
  - Facility #1, Melbourne
  - Facility #1, Randwick
- China (22):
  - Facility #1, Beijing, Beijing Municipality
  - Facility #1, Chongqing, Chongqing Municipality
  - Facility #1, Xiamen, Fujian
  - Facility #1, Guangzhou, Guangdong
  - Facility #2, Guangzhou, Guangdong
  - Facility #1, Harbin, Heilongjiang
  - Facility #1, Changchun, Jilin
  - Facility #1, Xi'an, Shaanxi
  - Facility #2, Xi'an, Shaanxi
  - Facility #3, Xi'an, Shaanxi
  - Facility #1, Taiyuan, Shan'xi
  - Facility #1, Jinan, Shandong
  - Facility #2, Jinan, Shandong
  - Facility #1, Qingdao, Shandong
  - Facility #1, Shanghai, Shanghai Municipality
  - Facility #2, Shanghai, Shanghai Municipality
  - Facility #3, Shanghai, Shanghai Municipality
  - Facility #1, Chengdu, Sichuan
  - Facility #2, Chengdu, Sichuan
  - Facility #1, Tianjin, Tianjin Municipality
  - Facility #1, Kunming, Yunnan
  - Facility #1, Wenzhou, Zhejiang
- Japan (60):
  - Eisai Trial Site #1, Nagoya, Aichi-ken
  - Eisai Trial Site #2, Nagoya, Aichi-ken
  - Eisai Trial Site #3, Nagoya, Aichi-ken
  - Eisai Trial Site #1, Tōon, Ehime
  - Eisai Trial Site #1, Yoshida-gun, Fukui
  - Eisai Trial Site #1, Kitakyushu, Fukuoka
  - Eisai Trial Site #1, Koga, Fukuoka
  - Eisai Trial Site #1, Kurume, Fukuoka
  - Eisai Trial Site #1, Sapporo, Hokkaido
  - Eisai Trial Site #2, Sapporo, Hokkaido
  - Eisai Trial Site #1, Itami, Hyōgo
  - Eisai Trial Site #1, Tsuchiura, Ibaraki
  - Eisai Trial Site #1, Kanazawa, Ishikawa-ken
  - Eisai Trial Site #1, Zentsujichó, Kagawa-ken
  - Eisai Trial Site #1, Fujisawa, Kanagawa
  - Eisai Trial Site #1, Kawasaki, Kanagawa
  - Eisai Trial Site #1, Gōshi, Kumamoto
  - Eisai Trial Site #1, Tamana, Kumamoto
  - Eisai Trial Site #1, Iwanuma, Miyagi
  - Eisai Trial Site #1, Sendai, Miyagi
  - Eisai Trial Site #1, Miyakonojō, Miyazaki
  - Eisai Trial Site #1, Ōmura, Nagasaki
  - Eisai Trial Site #1, Beppu, Oita Prefecture
  - Eisai Trial Site #1, Kurashiki, Okayama-ken
  - Eisai Trial Site #1, Izumi, Osaka
  - Eisai Trial Site #1, Sakai, Osaka
  - Eisai Trial Site #2, Sakai, Osaka
  - Eisai Trial Site #1, Sayama, Osaka
  - Eisai Trial Site #1, Takatsuki, Osaka
  - Eisai Trial Site #1, Asaka, Saitama
  - Eisai Trial Site #1, Higashimurayama, Saitama
  - Eisai Trial Site #1, Moriyama, Shiga
  - Eisai Trial Site #1, Matsue, Shimane
  - Eisai Trial Site #1, Hamamatsu, Shizuoka
  - Eisai Trial Site #1, Komatsushimachō, Tokushima
  - Eisai Trial Site #1, Kodaira, Tokyo
  - Eisai Trial Site #1, Kokubunji, Tokyo
  - Eisai Trial Site #1, Ube, Yamaguchi
  - Eisai Trial Site #1, Akita
  - Eisai Trial Site #1, Aomori
  - Eisai Trial Site #1, Fukui
  - Eisai Trial Site #1, Fukuoka
  - Eisai Trial Site #2, Fukuoka
  - Eisai Trial Site #1, Gifu
  - Eisai Trial Site #1, Hiroshima
  - Eisai Trial Site #2, Hiroshima
  - Eisai Trial Site #1, Kagoshima
  - Eisai Trial Site #2, Kagoshima
  - Eisai Trial Site #1, Kumamoto
  - Eisai Trial Site #1, Kyoto
  - Eisai Trial Site #1, Miyazaki
  - Eisai Trial Site #1, Nara
  - Eisai Trial Site #1, Niigata
  - Eisai Trial Site #1, Okayama
  - Eisai Trial Site #1, Saitama
  - Eisai Trial Site #2, Saitama
  - Eisai Trial Site #1, Shizuoka
  - Eisai Trial Site #2, Shizuoka
  - Eisai Trial Site #1, Toyama
  - Eisai Trial Site #1, Yamagata
- Malaysia (4):
  - Facility #1, Kuala Lumpur
  - Facility #1, Perak
  - Facility #1, Pulau Pinang
  - Facility #1, Terengganu
- South Korea (14):
  - Facility #1, Busan
  - Facility #2, Busan
  - Facility #1, Daegu
  - Facility #1, Daejeon
  - Facility #1, Gwangju
  - Facility #1, Incheon
  - Facility #1, Seoul
  - Facility #2, Seoul
  - Facility #3, Seoul
  - Facility #4, Seoul
  - Facility #5, Seoul
  - Facility #6, Seoul
  - Facility #7, Seoul
  - Facility #8, Seoul
- Taiwan (5):
  - Facility #1, Taichung
  - Facility #1, Tainan
  - Facility #1, Taipei
  - Facility #2, Taipei
  - Facility #1, Taoyuan District
- Thailand (5):
  - Facility #1, Rajathevee
  - Facility #1, Tha Muang
  - Facility #2, Tha Muang
  - Facility #3, Tha Muang
  - Facility #4, Tha Muang

REFERENCES:
- [Derived] Bresnahan R, Hill RA, Wang J. Perampanel add-on for drug-resistant focal epilepsy. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD010961. doi: 10.1002/14651858.CD010961.pub2. PMID 37059702
- [Derived] Nishida T, Lee SK, Inoue Y, Saeki K, Ishikawa K, Kaneko S. Adjunctive perampanel in partial-onset seizures: Asia-Pacific, randomized phase III study. Acta Neurol Scand. 2018 Apr;137(4):392-399. doi: 10.1111/ane.12883. Epub 2017 Dec 17. PMID 29250772

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 119 investigative sites in Australia, China, Korea, Japan, Malaysia, Taiwan, and Thailand from 15th May 2012 to 28th May 2020. A total of 940 participants were enrolled and screened, of which 230 participants were screen failures, 710 participants were randomized and 707 participants were treated in this study.
Pre-assignment Details: This study included Core and Extension Phase. Core Phase consisted of 2 phases: Prerandomization (Baseline) and Randomization (Titration, Maintenance Period). Extension Phase consisted of 3 periods: Preconversion, Conversion, Maintenance Period. Participants received varying doses depending on which dose level they were assigned to in Core Phase and their individual tolerance but in Extension Phase, all participants were up-titrated to single target dose level of 12 milligram (mg) per day.
Groups:
- Core Phase: Placebo; Extension Phase: up to 12 mg Perampanel: Participants received perampanel-matched placebo tablets (6 tablets), orally, once daily before bedtime from Week 0 up to Week 18 (up to 19 weeks) in the Core Phase. Participants received placebo in Extension Phase as they received in Core Phase, orally, once daily before bedtime from Week 19 to Week 22 (preconversion period). Participants started receiving perampanel 2 mg tablet, orally, once daily which was then titrated as 2 mg weekly increments up to a maximum dose of 12 mg, orally, once daily up to Week 28 (conversion period). All participants could have their dose down or up titrated until an optimal dose was reached. After the conversion period, participants entered a maintenance period in which they received the perampanel dose orally, once daily, that provided the optimal combination of efficacy and tolerability before bedtime up to Week 75 or longer depending on the requirements of each country in the Extension Phase.
- Core Phase: Perampanel 4 mg; Extension Phase: up to 12 mg Perampanel: Participants received perampanel 2 mg tablet, orally, once daily before bedtime in Week 0 and then titrated up to maximum dose of 4 mg orally, once daily from Week 1 up to Week 5 (titration period), followed by perampanel 4 mg, orally, once daily from Week 6 up to Week 18 (maintenance period) in the Core Phase. Total duration of titration and maintenance period in Core Phase was 19 weeks. Participants received the same dose of perampanel 4 mg in Extension Phase as they received in Core Phase, orally, once daily before bedtime from Week 19 to Week 22 (preconversion period). Participants started receiving perampanel 4 mg tablet, orally, once daily which was then titrated as 2 mg weekly increments up to a maximum dose of 12 mg, orally, once daily up to Week 28 (conversion period). All participants could have their dose down or up titrated until an optimal dose was reached. After the conversion period, participants entered a maintenance period in which they received the perampanel dose orally, once daily, that provided the optimal combination of efficacy and tolerability before bedtime up to Week 75 or longer depending on the requirements of each country in the Extension Phase.
- Core Phase: Perampanel 8 mg; Extension Phase: up to 12 mg Perampanel: Participants received perampanel 2 mg tablet, orally, once daily before bedtime in Week 0 and then titrated up to maximum dose of 8 mg (weekly increment of 2 mg from Week 1 up to Week 3) orally, once daily for up to Week 5 (titration period), followed by perampanel 8 mg, orally, once daily from Week 6 up to Week 18 (maintenance period) in the Core Phase. Total duration of titration and maintenance period was 19 weeks in the Core Phase. Participants received the same dose of perampanel 8 mg in the Extension Phase as they received in Core Phase, orally, once daily before bedtime from Week 19 to Week 22 (preconversion period). Participants started receiving perampanel 8 mg tablet, orally, once daily which was then titrated as 2 mg weekly increments up to a maximum dose of 12 mg, orally, once daily up to Week 28 (conversion period). All participants could have their dose down or up titrated until an optimal dose was reached. After the conversion period, participants entered a maintenance period in which they received the perampanel dose orally, once daily, that provided the optimal combination of efficacy and tolerability before bedtime up to Week 75 or longer depending on the requirements of each country in the Extension Phase.
- Core Phase/Extension Phase: up to 12 mg Perampanel: Participants received perampanel 2 mg tablet, orally, once daily before bedtime in Week 0 and then titrated up to maximum dose of 12 mg (weekly increment of 2 mg from Week 1 up to Week 5) orally, once daily for up to Week 5 (titration period), followed by perampanel 12 mg, orally, once daily from Week 6 up to Week 18 (maintenance period) in the Core Phase. Total duration of titration and maintenance period was 19 weeks in the Core Phase. Participants received the same dose of perampanel 12 mg in the Extension Phase as they received in Core Phase, orally, once daily before bedtime from Week 19 to Week 22 (preconversion period) and continued receiving perampanel 12 mg, orally, once daily up to Week 28 (conversion period). All participants could have their dose down or up titrated until an optimal dose was reached. After the conversion period, participants entered a maintenance period in which they received the perampanel dose orally, once daily, that provided the optimal combination of efficacy and tolerability before bedtime up to Week 75 or longer depending on the requirements of each country in the Extension Phase.
Period: Core Phase
Arm/Group | Core Phase: Placebo; Extension Phase: up to 12 mg Perampanel | Core Phase: Perampanel 4 mg; Extension Phase: up to 12 mg Perampanel | Core Phase: Perampanel 8 mg; Extension Phase: up to 12 mg Perampanel | Core Phase/Extension Phase: up to 12 mg Perampanel
Started | 177 | 176 | 177 | 180
Treated (Safety Analysis Set) | 176 | 176 | 175 | 180
Completed | 152 | 156 | 147 | 144
Not Completed | 25 | 20 | 30 | 36
Not completed — Adverse Event | 4 | 5 | 15 | 20
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 16 | 11 | 9 | 13
Not completed — Pregnancy | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 2 | 1 | 1
Not completed — Other than specified | 1 | 2 | 2 | 2
Not completed — Not treated | 1 | 0 | 2 | 0
Period: Extension Phase
Arm/Group | Core Phase: Placebo; Extension Phase: up to 12 mg Perampanel | Core Phase: Perampanel 4 mg; Extension Phase: up to 12 mg Perampanel | Core Phase: Perampanel 8 mg; Extension Phase: up to 12 mg Perampanel | Core Phase/Extension Phase: up to 12 mg Perampanel
Started | 151 (Participants who completed Core Phase and gave consent, entered the Extension Phase.) | 156 | 146 (Participants who completed Core Phase and gave consent, entered the Extension Phase.) | 143 (Participants who completed Core Phase and gave consent, entered the Extension Phase.)
Completed | 56 | 40 | 54 | 46
Not Completed | 95 | 116 | 92 | 97
Not completed — Lack of Efficacy | 17 | 33 | 26 | 24
Not completed — Pregnancy | 2 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 43 | 48 | 42 | 33
Not completed — Adverse Event | 18 | 16 | 9 | 20
Not completed — Lost to Follow-up | 2 | 1 | 1 | 1
Not completed — Other than specified | 13 | 18 | 13 | 18

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included all participants who signed informed consent, were randomized, received at least one dose of study medication, and had at least one post-dose safety assessment.
Groups:
- Core Phase: Placebo: Participants received perampanel-matched placebo tablets (6 tablets), orally, once daily before bedtime from Week 0 up to Week 18 (up to 19 weeks).
- Core Phase: Perampanel 4 mg: Participants received perampanel 2 mg tablet, orally once daily before bedtime in Week 0 and then titrated up to maximum dose of 4 mg orally once daily from Week 1 up to Week 5 (titration period), followed by perampanel 4 mg, orally once daily from Week 6 up to Week 18 (maintenance period). Total duration of titration and maintenance period is 19 weeks.
- Core Phase: Perampanel 8 mg: Participants received perampanel 2 mg tablet, orally once daily before bedtime in Week 0 and then titrated up to maximum dose of 8 mg (weekly increment of 2 mg from Week 1 up to Week 3) orally once daily for up to Week 5 (titration period), followed by perampanel 8 mg, orally once daily from Week 6 up to Week 18 (maintenance period). Total duration of titration and maintenance period is 19 weeks.
- Core Phase: Perampanel 12 mg: Participants received perampanel 2 mg tablet, orally once daily before bedtime in Week 0 and then titrated up to maximum dose of 12 mg (weekly increment of 2 mg from Week 1 up to Week 5) orally once daily for up to Week 5 (titration period), followed by perampanel 12 mg, orally once daily from Week 6 up to Week 18 (maintenance period). Total duration of titration and maintenance period is 19 weeks.
- Total: Total of all reporting groups
Arm/Group | Core Phase: Placebo | Core Phase: Perampanel 4 mg | Core Phase: Perampanel 8 mg | Core Phase: Perampanel 12 mg | Total
Number analyzed (Participants) | 176 | 176 | 175 | 180 | 707
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (13.21) | 33.1 (13.18) | 33.6 (14.11) | 32.3 (12.30) | 33.4 (13.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 94 | 84 | 93 | 361
  Male | 86 | 82 | 91 | 87 | 346
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 176 | 175 | 175 | 179 | 705
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 169 | 168 | 159 | 171 | 667
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 7 | 14 | 7 | 35
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Core Phase: Percent Change in Seizure Frequency (For All Partial Seizures) Per 28 Days in the Randomization Phase Relative to Pre-randomization Phase (Baseline)
Description: Seizure frequency was based on number of seizures per 28 days, calculated as the number of seizures over the entire time interval divided by the number of days in the interval and multiplied by 28. All partial seizure included simple partial seizures without motor signs, simple partial with motor signs, complex partial, and complex partial with secondary generalized seizures. A simple partial seizure takes place on one side of the brain. Usually, people experiencing a simple partial seizure do not lose consciousness or awareness. A complex partial seizure is a type of seizure that arises in one lobe of the brain, rather than the whole brain. The seizure affects people's awareness and may cause them to lose consciousness.
Time Frame: Baseline, Week 19
Population: Intent-to-treat (ITT) Analysis Set included all participants who signed informed consent, were randomized, received at least one dose of study medication, and had at least one postdose seizure frequency data.
Measure: Median (Full Range); unit: percent change
Groups:
- Placebo: Participants received perampanel-matched placebo tablets (6 tablets), orally, once daily before bedtime from Week 0 up to Week 18 (up to 19 weeks).
- Perampanel 4 mg: Participants received perampanel 2 mg tablet, orally once daily before bedtime in Week 0 and then titrated up to maximum dose of 4 mg orally once daily from Week 1 up to Week 5 (titration period), followed by perampanel 4 mg, orally once daily from Week 6 up to Week 18 (maintenance period). Total duration of titration and maintenance period is 19 weeks.
- Perampanel 8 mg: Participants received perampanel 2 mg tablet, orally once daily before bedtime in Week 0 and then titrated up to maximum dose of 8 mg (weekly increment of 2 mg from Week 1 up to Week 3) orally once daily for up to Week 5 (titration period), followed by perampanel 8 mg, orally once daily from Week 6 up to Week 18 (maintenance period). Total duration of titration and maintenance period is 19 weeks.
- Perampanel 12 mg: Participants received perampanel 2 mg tablet, orally once daily before bedtime in Week 0 and then titrated up to maximum dose of 12 mg (weekly increment of 2 mg from Week 1 up to Week 5) orally once daily for up to Week 5 (titration period), followed by perampanel 12 mg, orally once daily from Week 6 up to Week 18 (maintenance period). Total duration of titration and maintenance period is 19 weeks.
Arm/Group | Placebo | Perampanel 4 mg | Perampanel 8 mg | Perampanel 12 mg
Number analyzed (Participants) | 175 | 174 | 175 | 180
percent change | -10.76 [-90.4 to 400.0] | -17.32 [-97.1 to 473.4] | -28.95 [-100.0 to 809.4] | -38.03 [-100.0 to 456.8]
Statistical Analysis 1: Comparison: Placebo vs Perampanel 4 mg; Test type: Superiority; p = 0.2330, ANCOVA; Median Difference (Final Values) = -5.09, 95% CI 2-sided [-14.112 to 4.519] — Median Difference to placebo and the 95 percent (%) confidence interval are based on the Hodges-Lehmann method
Statistical Analysis 2: Comparison: Placebo vs Perampanel 8 mg; Test type: Superiority; p = 0.0003, ANCOVA; Median Difference (Final Values) = -16.45, 95% CI 2-sided [-25.683 to -7.251] — Median Difference to placebo and the 95% confidence interval are based on the Hodges-Lehmann method
Statistical Analysis 3: Comparison: Placebo vs Perampanel 12 mg; Test type: Superiority; p < 0.0001, ANCOVA; Median Difference (Final Values) = -24.95, 95% CI 2-sided [-33.878 to -16.235] — Median Difference to placebo and the 95% confidence interval are based on the Hodges-Lehmann method

2. Secondary Outcome: Core Phase: Responder Rate During the Maintenance Period of the Randomization Phase Relative to the Prerandomization Phase (Baseline)- Last Observation Carried Forward (LOCF)
Description: Responder rate was percentage of participants with greater than or equal to (>=) 50% reduction in seizure frequency during maintenance period of the randomization phase relative to prerandomization phase (baseline). If the reduction in seizure frequency is less than (<) 50%, then the participants are considered as non-responders.
Time Frame: Baseline, Week 19
Population: ITT Analysis Set included all participants who signed informed consent, were randomized, received at least one dose of study medication, and had at least one postdose seizure frequency data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Perampanel 4 mg | Perampanel 8 mg | Perampanel 12 mg
Number analyzed (Participants) | 175 | 174 | 175 | 180
percentage of participants | 19.4 | 23.0 | 36.0 | 43.3
Statistical Analysis 1: Comparison: Placebo vs Perampanel 4 mg; Test type: Superiority; p = 0.3954, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Perampanel 8 mg; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Perampanel 12 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Core Phase: Percent Change in Seizure Frequency Per 28 Days For Complex Partial Seizures Plus Secondary Generalized Seizures in the Randomization Phase Relative to the Prerandomization Phase (Baseline)
Description: Seizure frequency was based on number of seizures per 28 days, calculated as the number of seizures over the entire time interval divided by the number of days in the interval and multiplied by 28. A complex partial seizure is a type of seizure that arises in one lobe of the brain, rather than the whole brain and it affects awareness and may cause in loss of consciousness. Secondary generalized seizures begin in one part of the brain, but then spread to both sides of the brain.
Time Frame: Baseline, Week 19
Population: ITT Analysis Set included all participants who signed informed consent, were randomized, received at least one dose of study medication, and had at least one postdose seizure frequency data. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Perampanel 4 mg | Perampanel 8 mg | Perampanel 12 mg
Number analyzed (Participants) | 158 | 151 | 157 | 167
percent change | -11.70 [-88.6 to 400.0] | -19.08 [-100.0 to 410.0] | -33.68 [-100.0 to 1103.4] | -41.80 [-100.0 to 456.8]
Statistical Analysis 1: Comparison: Placebo vs Perampanel 4 mg; Test type: Superiority; p = 0.0552, ANCOVA; Median Difference (Final Values) = -8.27, 95% CI 2-sided [-18.067 to 1.671] — Median Difference to placebo and the 95% confidence interval are based on the Hodges-Lehmann method
Statistical Analysis 2: Comparison: Placebo vs Perampanel 8 mg; Test type: Superiority; p < 0.0001, ANCOVA; Median Difference (Final Values) = -21.21, 95% CI 2-sided [-30.941 to -11.368] — Median Difference to placebo and the 95% confidence interval are based on the Hodges-Lehmann method
Statistical Analysis 3: Comparison: Placebo vs Perampanel 12 mg; Test type: Superiority; p < 0.0001, ANCOVA; Median Difference (Final Values) = -28.65, 95% CI 2-sided [-37.698 to -19.794] — Median Difference to placebo and the 95% confidence interval are based on the Hodges-Lehmann method

4. Secondary Outcome: Core Phase: Number of Participants With Clinical Global Impression of Change (CGIC) Scores
Description: The investigator evaluated each participant for CGIC questionnaire to assess change in participant's disease clinical status from baseline. Assessment evaluated frequency of seizures, severity of seizures, occurrence of adverse events (AEs), and overall functional status of the participant using the 7-point scale. The evaluation used a 7-point scale with the scores 1: Very much improved, 2: Much improved, 3: Minimally improved, 4: No change, 5: Minimally worse, 6: Much worse, 7: Very much worse. Lower score indicated improvement and higher score indicated worsening.
Time Frame: Baseline, Week 19
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Perampanel 4 mg | Perampanel 8 mg | Perampanel 12 mg
Number analyzed (Participants) | 175 | 174 | 175 | 180
Participants
  Very much improved | 3 | 5 | 11 | 9
  Much improved | 31 | 39 | 41 | 54
  Minimally improved | 54 | 45 | 53 | 40
  No change | 67 | 56 | 37 | 37
  Minimally worse | 3 | 10 | 5 | 4
  Much worse | 1 | 0 | 0 | 1
  Very much worse | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From the date of first dose up to 30 days after the last dose of study drug (up to Week 79)
Description: Planned safety analysis of Extension Phase included treatment emergent AEs on/after first day of perampanel treatment in entire study. Analysis set for Extension Phase included 679 participants: 596 had perampanel in Core Phase & at least one dose of perampanel in Extension Phase, 83 had perampanel in Core Phase only. Participants received varying doses in Extension Phase depending on tolerance but as target dose was defined as 12 mg/day for all participants, AEs were summarized as a single arm.
Groups:
- Extension Phase: Perampanel 12 mg: Participants received the same dose of perampanel in Extension Phase as they received in Core Phase, orally, once daily before bedtime from Week 19 to Week 22 (preconversion period). This dose was then titrated as 2 mg weekly increments up to a maximum dose of 12 mg, orally once daily up to Week 28 (conversion period). Participants who received perampanel matched-placebo in Core Phase were given perampanel 2 mg weekly increments up to a maximum dose of 12 mg, orally once daily up to Week 28 (conversion period). All participants were allowed to have their dose down or up titrated until an optimal dose was reached. A maintenance period was followed by conversion period in which participants received perampanel dose of 12 mg, orally, once daily, that provided the optimal combination of efficacy and tolerability before bedtime up to Week 75 or longer depending on the requirements of each country.
Arm/Group | Core Phase: Placebo | Core Phase: Perampanel 4 mg | Core Phase: Perampanel 8 mg | Core Phase: Perampanel 12 mg | Extension Phase: Perampanel 12 mg
All-Cause Mortality (participants affected / at risk) | 1/176 | 0/176 | 1/175 | 0/180 | 7/679
Serious Adverse Events (participants affected / at risk) | 10/176 | 6/176 | 7/175 | 12/180 | 113/679
Other Adverse Events (participants affected / at risk) | 114/176 | 119/176 | 127/175 | 155/180 | 618/679
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Phase: Placebo (N=176) | Core Phase: Perampanel 4 mg (N=176) | Core Phase: Perampanel 8 mg (N=175) | Core Phase: Perampanel 12 mg (N=180) | Extension Phase: Perampanel 12 mg (N=679)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Renal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (7)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 6 (6)
Complex partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Partial seizures with secondary generalisation (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (4)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Acute psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conversion disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Self-injurious ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sudden unexplained death in epilepsy (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Emotional disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postictal psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Psychogenic seizure (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Focal dyscognitive seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Idiopathic partial epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limbic encephalitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Seizure cluster (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Lens dislocation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival hypertrophy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Phase: Placebo (N=176) | Core Phase: Perampanel 4 mg (N=176) | Core Phase: Perampanel 8 mg (N=175) | Core Phase: Perampanel 12 mg (N=180) | Extension Phase: Perampanel 12 mg (N=679)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 12 (13)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 3 (3) | 5 (6) | 4 (4) | 23 (25)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 12 (13)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 11 (12)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (6)
Dysmetropsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Keratoconjunctivitis sicca (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Normal tension glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Retinal disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (4) | 4 (4) | 10 (10) | 35 (37)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 3 (3) | 4 (4) | 6 (6) | 33 (42)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 2 (2) | 5 (6) | 3 (3) | 25 (35)
Constipation (Gastrointestinal disorders) | 1 (2) | 2 (2) | 5 (5) | 1 (1) | 27 (36)
Vomiting (Gastrointestinal disorders) | 7 (8) | 1 (1) | 1 (1) | 3 (3) | 24 (25)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 11 (13)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 13 (15)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 11 (11)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 7 (7)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 10 (10)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (4)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 23 (25)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 8 (8)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gingival hyperplasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gingival ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis atrophic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Irritability (General disorders) | 1 (1) | 8 (9) | 10 (10) | 9 (9) | 0 (0)
Fatigue (General disorders) | 5 (5) | 4 (4) | 6 (6) | 9 (9) | 34 (36)
Gait disturbance (General disorders) | 3 (3) | 2 (2) | 4 (4) | 9 (9) | 28 (34)
Pyrexia (General disorders) | 3 (6) | 2 (2) | 4 (4) | 4 (6) | 39 (90)
Asthenia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 17 (20)
Malaise (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 5 (5)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (7)
Device breakage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Foreign body reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (9)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 6 (6)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Nasopharyngitis (Infections and infestations) | 26 (26) | 23 (23) | 24 (30) | 23 (28) | 170 (325)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 8 (12) | 14 (17) | 11 (19) | 70 (147)
Pharyngitis (Infections and infestations) | 3 (3) | 1 (2) | 4 (5) | 2 (2) | 24 (36)
Influenza (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 31 (36)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 18 (20)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 8 (9)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 7 (7)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 12 (13)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (10)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
Purulence (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Syphilis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (8)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 8 (10)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eczema infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (5) | 5 (19) | 6 (6) | 5 (5) | 49 (81)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1) | 2 (4) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 12 (13)
Skin laceration (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 21 (21)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 14 (15)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 8 (9)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 14 (20)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 11 (13)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 8 (8)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 5 (5)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (3)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Weight increased (Investigations) | 1 (1) | 7 (8) | 6 (6) | 6 (6) | 40 (44)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (2) | 2 (2) | 5 (5) | 24 (32)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 9 (13)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 9 (10)
Protein urine present (Investigations) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 12 (14)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 13 (14)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Blood uric acid increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 7 (7)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood parathyroid hormone abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6)
Blood triglycerides abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Monocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Red blood cells urine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine ketone body present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood urine present (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 5 (5) | 3 (3) | 21 (21)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 10 (12)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 6 (6)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 6 (6)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 7 (8)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Weight fluctuation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Appetite disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 20 (22)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 10 (13)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 9 (9)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 14 (15)
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Myokymia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 10 (11) | 40 (48) | 50 (60) | 76 (85) | 317 (435)
Somnolence (Nervous system disorders) | 23 (24) | 28 (28) | 31 (36) | 32 (33) | 165 (199)
Headache (Nervous system disorders) | 13 (18) | 12 (22) | 13 (14) | 10 (11) | 94 (164)
Ataxia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 7 (8) | 22 (26)
Balance disorder (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1) | 4 (4) | 17 (18)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (4) | 22 (24)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 3 (4) | 1 (1) | 2 (2) | 12 (17)
Tremor (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 19 (23)
Convulsion (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 14 (16)
Nystagmus (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Amnesia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 9 (9)
Complex partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 6 (6)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 3 (5)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Clumsiness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cranial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 5 (7)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nerve root compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyslalia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Partial seizures with secondary generalisation (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Tongue biting (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aggression (Psychiatric disorders) | 0 (0) | 4 (4) | 5 (5) | 4 (4) | 22 (24)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 3 (3) | 7 (7) | 2 (2) | 21 (28)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 6 (6) | 1 (1) | 22 (22)
Insomnia (Psychiatric disorders) | 7 (7) | 3 (4) | 2 (2) | 3 (3) | 25 (27)
Mood swings (Psychiatric disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 12 (13)
Anger (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 9 (9)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 16 (19)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 6 (6)
Depressed mood (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Sleep disorder (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 7 (8)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Confusional arousal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Emotional disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Expressive language disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fear (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Impatience (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Personality disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Regressive behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Self-injurious ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sleep talking (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Soliloquy (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stubbornness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
Thinking abnormal (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tic (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute stress disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Bladder irritation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nocturia (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Cervical cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypomenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6)
Pelvic fluid collection (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 13 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 8 (10)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 5 (10)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (6)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 9 (11)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 9 (9) | 31 (37)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 13 (16)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 18 (20)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 13 (13)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 1 (1) | 2 (2) | 8 (9)
Heat rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (9)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 6 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pityriasis alba (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Angiodysplasia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chemical poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Closed globe injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear canal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eyelid contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 23 (24)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 16 (18)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anticonvulsant drug level increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood magnesium abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood sodium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroxine free decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
pH urine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Change in seizure presentation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysstasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Focal dyscognitive seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyposmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Language disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postictal headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postural tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radial nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 16 (19)
Seizure cluster (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Sleep deficit (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Slow response to stimuli (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonic convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Borderline glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Corneal erosion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excessive eye blinking (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid myoclonus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Psychogenic visual disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Xerophthalmia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Breath odour (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Gingival hypertrophy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Noninfective gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral contusion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary gland mucocoele (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ketonuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Androgenetic alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture blisters (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Product blister packaging issue (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angular cheilitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bartholin's abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carbuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (12)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dermatophytosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eczema impetiginous (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Gingival abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes dermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mumps (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pericoronitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea manuum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Benign hepatobiliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hearing aid user (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Decreased activity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruxism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Conversion disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dissociative disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enuresis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impulsive behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Middle insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Persecutory delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Persistent depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychogenic seizure (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Somatic symptom disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menstruation delayed (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oligomenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scrotal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 61 (72)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes